CLINICAL TRIAL: NCT01658072
Title: Analgesia After Total Hip Arthroplasty: Peri-Articular Injection Versus Epidural Patient Controlled Analgesia
Brief Title: Analgesia After Total Hip Arthroplasty: Peri-Articular Injection Versus Epidural Patient Controlled Analgesia (PCA)
Acronym: PAI Hip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-053
Record Dates: First submitted 2012-03-01; First posted 2012-08-06 (Estimated); Results first posted 2016-05-10 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis
Keywords: Total Hip Arthroplasty; Total Hip Replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peri-Articular Injection (Experimental)
  Interventions: Procedure: Peri-Articular Injection
- Epidural Patient Controlled Analgesia (Epidural PCA) (Active Comparator)
  Interventions: Procedure: Epidural Patient Controlled Analgesia (Epidural PCA)

INTERVENTIONS:
Procedure: Peri-Articular Injection — Use of a different analgesic protocol, based on a peri-articular injection
  Arms: Peri-Articular Injection
Procedure: Epidural Patient Controlled Analgesia (Epidural PCA) — Epidural analgesia pathway.
  Arms: Epidural Patient Controlled Analgesia (Epidural PCA)

SUMMARY:
The best way to provide analgesia after total hip arthroplasty is hotly debated. There are two protocols in use at Hospital for Special Surgery(HSS). Both protocols have their proponents, but there are limited data for making an informed choice of protocols. For total hip arthroplasty at HSS, epidural analgesia is used most frequently as it reduces pain with physical therapy. However, epidural analgesia can be associated with nausea, pruritis, dizziness, and orthostatic hypotension. These side-effects can slow physical therapy and may prolong the time until the patient is ready for discharge. Some surgeons at HSS have decided to use a different analgesic protocol, based on a peri-articular injection. This protocol avoids epidural analgesia and systemic opioids. However, patients are given oral opioids as part of a multimodal pain therapy. The investigators propose to compare peri-articular injection to epidural patient controlled analgesia (Epidural PCA). The investigators will enroll 90 total patients (45 per study arm). The enrollment period will be approximately one year and the duration of the follow-up with study patients will be three months following their procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis scheduled for primary total hip arthroplasty with a participating surgeon
* Age 50 to 80 years old
* Planned use of regional anesthesia
* Ability to follow study protocol

Exclusion Criteria:

* Patients younger than 50 years old and older than 80
* Patients intending to receive general anesthesia
* Allergy or intolerance to one of the study medications
* Patients with an ASA of IV
* Patients with insulin-dependent diabetes
* Patients with hepatic (liver) failure
* Patients with chronic renal (kidney) failure
* Chronic opioid use (taking opioids for longer than 3 months)
* Patients with any prior major ipsilateral hip surgery
* Allergy to any of the medications (or adhesives) involved in the protocol

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kethy M Jules-Elysee, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peri-Articular Injection | Epidural Patient Controlled Analgesia (Epidural PCA)
Started | 45 | 45
Completed | 41 | 43
Not Completed | 4 | 2
Not completed — Protocol Violation | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peri-Articular Injection | Epidural Patient Controlled Analgesia (Epidural PCA) | Total
Number analyzed (Participants) | 41 | 43 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.5) | 64.8 (7.1) | 64.3 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 20 | 24 | 44
Region of Enrollment [Number; unit: participants]
  United States | 41 | 43 | 84
Body mass index [Mean (Standard Deviation); unit: kg/(m^2)] | 28.0 (5.4) | 27.9 (6.2) | 28.0 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Time Until Patient is Ready for Discharge
Description: "readiness for discharge" to home or to a rehabilitation facility (compared to the HSS standard regimen of epidural analgesia) after total hip arthroplasty.
Time Frame: Length of Hospital Stay, an expected average of 3 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Peri-Articular Injection | Epidural Patient Controlled Analgesia (Epidural PCA)
Number analyzed (Participants) | 41 | 43
days | 2.4 (0.7) | 2.3 (0.8)

ADVERSE EVENTS:
Arm/Group | Peri-Articular Injection | Epidural Patient Controlled Analgesia (Epidural PCA)
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes